CLINICAL TRIAL: NCT07131969
Title: Transcriptional Analysis of Mechanisms and Predictors in Acute Liver Failure and Sepsis
Brief Title: Transcriptional Analysis of Mechanisms in Liver Failure and Sepsis
Acronym: MAP-ALF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Dhupal Patel, Principal investigator, University of Cambridge
Other Study IDs: A097365
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acute Liver Failure; Sepsis
Keywords: acute liver failure; sepsis; transcriptional analysis; predictors; paracetamol overdose; acetaminophen overdose
MeSH Terms: conditions — Liver Failure, Acute; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood collected in Tempus tubes for RNA-sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute liver failure or sepsis
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — Venous blood sampling into Tempus tube for RNA-sequencing

SUMMARY:
Context Acute liver failure (ALF) is a life-threatening condition that occurs on the background of a healthy liver. The most common cause of acute liver failure in the UK is paracetamol overdose. Acute liver failure results from liver damage and activation of the body's inflammatory defences with subsequent damage to other organs including kidneys, lungs and heart. This often requires life support in an intensive care unit before liver transplantation (LT), the only currently available and effective rescue treatment for acute liver failure.

Challenge Patient factors and organ availability limit who can benefit from liver transplant. At present there are no effective alternative therapies for patients who do not get a liver transplant, and survival rates in these situations are poor. The underlying mechanisms of inflammation are poorly understood, thus therapies are limited.

Aim The investigators research aims to understand the mechanisms that underpin the inflammation seen in acute liver failure by studying the inflammatory cells in the blood and examining their cellular programmes. This will allow the investigators to identify pathways that are activated and understand how the liver and blood interact to spread inflammation around the body. The investigators aim to identify targets for disease-modifying therapies to avert the need for liver transplant.

Importance Understanding how the body responds to acute liver failure, and whether there are different patterns of inflammatory response, will enable trials of immune-modulating drugs to prevent the need for liver transplantation or prolong the time a patient can wait for an organ. This has the potential to help improve organ availability for other patients and save lives in acute liver failure.

ELIGIBILITY:
Inclusion Criteria:

* acute liver failure due to acetaminophen (paracetamol) overdose admitted to ICU
* all cause sepsis admitted to ICU

Exclusion Criteria:

* age <16y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute liver failure due to acetaminophen overdose OR sepsis who are admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | From enrolment until at least 1-year

SECONDARY OUTCOMES:
Transplant free survival | From enrolment to at least one year
  30-day and 1-year survival without transplant
Length of stay - ICU and hospital | From enrolment
  Number of days stayed in ICU and in-hospital
Transplant free mortality | From enrolment until death (at least until 1year)
  Death without transplant

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - University Hospitals Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - Leeds General Infirmary, Leeds
  - Kings College Hospital, London
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: Undecided